CLINICAL TRIAL: NCT05225077
Title: Effect of Short-term Dapagliflozin on Renal Function After Heart Catheterization or Percutaneous Coronary Intervention in Patients With Chronic Kidney Disease
Brief Title: Short-term Use of Dapagliflozin to Protect Kidney Function in CKD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, Professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROTECT-CKD
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Renal Insufficiency, Chronic; Cardiac Catheterization; Percutaneous Coronary Intervention
Keywords: Sodium-Glucose Transporter 2 Inhibitors; Dapaglifozin; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10mg group (Active Comparator): Dapagliflozin 10 mg once a day for 1 month after the procedure.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]
- Non-intervention group (No Intervention): No intervention.

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Dapagliflozin 10 mg once a day for 1 month after CAG or PCI.
  Arms: Dapagliflozin 10mg group

SUMMARY:
This study aim to investigate the protected effects of short-term use of dapagliflozin (administered within 3 days after procedure) in CKD patients after coronary angiography or percutaneous coronary intervention, as well as observed the incidence of CIN.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Written informed consent
* Glomerular Filtration Rate (GFR)≥ 30 ml/min/1.73m2 [CKD stage G1-G3]
* Percutaneous coronary intervention in patients with NSTEMI, UA, STCD and asymptomatic patients

Exclusion Criteria:

* Active malignancy
* Class I or equivalent indication for treatment with a SGLT2 inhibitor
* Pregnancy or willing of pregnancy during the follow up period
* Active urogenital infection
* Diabetes mellitus type 1
* History of diabetic ketoacidosis
* Cardiogenic shock
* eGFR < 29 ml/min/1.73m2

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast induced nephropathy | 48 hours
  Serum creatinine (Scr) elevation of >25% or >0.5 mg/dl (44 μmol/l) from baseline within 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dong A University Hospital, Busan, South Korea